CLINICAL TRIAL: NCT00388180
Title: A Randomized, Double-blind, Parallel Group Study to Evaluate the Effect of 12-week Treatment With GW590735X (20ug) or GW501516X (10mg) Relative to Placebo on Measures of Adiposity and Inflammation in Overweight and Obese Subjects
Brief Title: An Exploratory Study To Look At The Effect Of Two Investigational Drugs On Body Fat And Inflammation
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: PAD100958
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Hypercholesterolemia; Dyslipidaemias; Obesity
Keywords: cholesterol; inflammation; fat
MeSH Terms: conditions — Hypercholesterolemia; Obesity; Inflammation; Platelet Glycoprotein IV Deficiency | interventions — GW 501516; 2-methyl-2-(4-(((4-methyl-2-(4-trifluoromethylphenyl)-thiazol-5-ylcarbonyl)amino)methyl)phenoxy)propionic acid

INTERVENTIONS:
Drug: GW501516
Drug: GW590735
  Other Names: GW501516

SUMMARY:
The investigational drugs administered in this study activate proteins called PPARs. Data in the scientific literature on PPARs, as well as animal data and early clinical data generated by GSK with these drugs, suggest that activation of PPARs may cause the body to increase its use of fatty acids for energy, and lead to a reduction in body fat. There are also data to suggest a role for PPARs in regulating lipid (e.g., cholesterol) levels and inflammation. These and other activities of PPARs are being further explored in this clinical study.

ELIGIBILITY:
Inclusion criteria:

* Body Mass Index in the range of 27 - 43 kg/m2
* Waist circumference > 95cm

Exclusion criteria:

* Clinically relevant abnormalities on screening ECG/holter, labs or medical examination
* Use of tobacco within 6 months of the study
* Regular strenuous exercise
* Use of prescription or non-prescription medications, including vitamins and herbal/dietary supplements
* LDL < 80mg/dL; TG <100mg/dL or >400mg/dL

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2004-12

PRIMARY OUTCOMES:
Body fat levels

SECONDARY OUTCOMES:
Levels of multiple proteins/biomarkers in blood and fat tissue, as well as specific lipid in muscle and liver (via imaging). Gene expression in blood and fat tissue.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Olson EJ, Pearce GL, Jones NP, Sprecher DL. Lipid effects of peroxisome proliferator-activated receptor-delta agonist GW501516 in subjects with low high-density lipoprotein cholesterol: characteristics of metabolic syndrome. Arterioscler Thromb Vasc Biol. 2012 Sep;32(9):2289-94. doi: 10.1161/ATVBAHA.112.247890. Epub 2012 Jul 19. PMID 22814748